CLINICAL TRIAL: NCT02068118
Title: Optimisation de la Surveillance Ambulatoire Des Insuffisants CArdiaques Par Télécardiologie (OSICAT)
Brief Title: Optimization of the Ambulatory Monitoring for Patients With Heart Failure by Tele-cardiology
Acronym: OSICAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CDM e-Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-A01672-41
Record Dates: First submitted 2014-02-17; First posted 2014-02-21 (Estimated); Results first posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-09

CONDITIONS: Chronic Heart Failure
Keywords: E health; Telemonitoring; Prevention; Heart Failure; Cordiva; Telecardiology Program; Remote Patient Management; Education
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (No Intervention): Standard follow-up, with conventional monitoring involving consultations and monitoring by their general practitioners or referring cardiologists
- Tele-cardiology group (Experimental): Telecardiology Program
  Interventions: Device: Telecardiology program

INTERVENTIONS:
Device: Telecardiology program — The telecardiology program is a combination of a scale, a device asking the patients questions about the symptoms associated with their heart failure, and regular phone calls made by nurses.
  Automatic algorithms have been built-up in order to detect early the need for a hospitalization due to heart failure.
  Arms: Tele-cardiology group

SUMMARY:
Targeted population: Patients with heart failure causing hospitalization during the last twelve months.

Hypothesis: The number of all cause deaths and hospitalizations will be smaller for the Telecardiology group than for the reference group (standard follow-up care). An 18 months period of observation is required.

Main goal: To compare the rate of all cause deaths and hospitalizations of patients with heart failure between the Telecardiology group and the reference group after 18 months of monitoring.

DETAILED DESCRIPTION:
COMPARATIVE STUDY:

Comparative study of patients with chronic heart failure, randomized ratio (1:1), with two study arms (telecardiology vs usual care). French multicenter study.

The planned enrolment is 990 patients in a total period of 3.5 years. This study will involve an enrolment visit, managed by the recruiting investigator cardiologist, then four telephone contacts by Clinical Studies Technicians (CST). The purpose of the CST telephone contacts is to record the study data, and this will be occur for both study arms. Throughout the study, the patients in the telecardiology study arm will have regular contact with the Cordiva nurses for the management of their chronic heart failure, through telemonitoring and coaching. There is no planned hospitalization for the study.

Patients in the control group will receive the usual care: After enrolment, they will return home and will subsequently have regular visits to their General Practitioner (GP) or referring cardiologist.

Patients in the telecardiology group will receive the necessary monitoring equipment in their home in the week following their enrolment visit. This equipment includes a connected electronic scale and a questionnaire box. This questionnaire is designed to evaluate the evolution of patient symptoms.

During the presentation of the study to the patient before study inclusion, the investigator will inform the patient about the use of the equipment.

The material provided is "self installable" but if the patient asks for help, the equipment will be installed at the patient's home by a private nurse, who also will check that the patient knows how to use the equipment.

Each patient will respond daily to 8 yes/no questions:

* Did you have more breathing issues last night than the previous night?
* Did you need an extra pillow for better breathing last night?
* Do you cough more than usual?
* Are your legs are more swollen than usual?
* Do you feel yourself more tired than usual?
* Have you had or do you have a fever above 38.5 °C?
* Have you felt or do you feel palpitations?
* Do you find that your physical activity is more limited today than the previous days?

Patients should simply answer yes or no to all of these questions through the questionnaire box.

The self-monitoring parameters (weight and questionnaire answers) will be remotely transmitted via standard phone lines (wired, 3G or GPRS) to the secured servers.

These data will be analyzed automatically by an expert system that will generate an alert in case of abnormal values. The objective is to anticipate possible acute cardiac failure.

The specialized nurses from the Cordiva center will manage those alerts during working hours and will contact the patient to validate with him the relevance of the alert. If the clinical reality of the alert is confirmed, the nurse will advise the patient to contact his GP or referring cardiologist. In parallel to the nurse advising the patient, the referring physician will receive an alert report including the weight values and the symptoms which triggered this alert. Then, he can then take any action he considers appropriate.

A binder will be sent to the patients. This will contain various information related to the management of their heart failure: heart physiology, symptoms, treatments, diet, physical activity...

The purpose of this binder is to support the discussion between the Cordiva nurses and the patient.

Upon receipt and installation of the equipment in the patient's home, the nurses will arrange a first telephone interview, which will last approximately 45 minutes. The nurses will first introduce the team and the overall clinical approach, and will have a discussion with the patient to better understand the patient (anamnesis, treatment, psycho-social profile, smoking, alcohol use, physical activity, and so on).

After this call, patient and nurse will together determine together the date for the next phone call date.

On a regular basis (for example every three weeks), a Cordiva nurse will call the patient to check the current status of his disease and its treatment, and to assist him in the management of his disease on a daily basis (compliance, physical activity, nutrition, illness experience... ) . This call will last approx. 15 minutes, however, the duration of the call is not limited, but is defined according to the needs of the patient.

At the end of each call, the nurse will define with the patient educational goals (disease knowledge, treatments, recognizing acute episodes symptoms, learning better health habits, practise regular physical activity).

Cordiva center is also available for patient's inbound calls. In this way, patients will be able to easily call the center during working hours, and discuss with a specialized Cordiva nurse. This line is not an emergency line and does not replace the 112, which remains the only accredited contact in case of emergencies.

In case of temporary travel of the patient away from home (i.e. for holidays), the patient can take the box and scale with him. This material is provided with GPRS SIM card, so the connection will be maintained. The patient may also provide an alternative phone number for the calls with the nurses.

The patient's GP will be involved in this outpatient care from the beginning of the study. Indeed, data collected through the connected boxes and scales will be displayed in dedicated reports sent to the GP. These reports will be transmitted every 2 months. These reports will also be sent to the referring cardiologist if requested.

Moreover, in case of validated alerts, the referring physician will have access to a weight and symptoms report, allowing him to take any action he thinks appropriate.

ABOUT CORDIVA CENTER: The center has a team of specialized and graduated nurses in heart failure management and in therapeutic education, due to the dedicated training they have received. Indeed, many studies in the multidisciplinary care of heart failure patients have demonstrated the key role of nurses, acting as bridge between patients and health professionals.

The nurses take care of patient compliance based on the referring cardiologist or general practitioner instructions, and monitor patient clinical parameters (weight and symptoms). The nurses use a software based interviews guide. Patient objectives are defined based on information regarding certain factors (health status, clinical signs, drugs), and this information will be collected by the nurses into a computerized database. This information is requested in strict patient accompanying perspective and therefore do not appear in the study results.

The two data sets (data collected by nurses for patient management on one hand, and data collected by CST for the study on another hand) will never be connected and only study data from CST will be used to assess study criteria.

To evaluate patient knowledge and needs, the nurses use active listening (open questions, paraphrasing, empathy and positive reinforcement). These techniques help them to customize information and messages and reinforce personalized care. Cordiva center nurses benefit from specialized training in motivational interviewing. They have also received dedicated training in cardiology and heart failure, "mental state" of heart failure patients, communication and patient education.

Coherence of this informative approach is guaranteed on one hand because of the tools available for the nurses (binder, interview guide), and on the other hand because of the center organization itself: monitoring of patients insured by team of nurses, weekly debrief of recorded calls…

EXTENSION PERIOD:

The extension period will be conducted on an open, non-comparative basis. The aim of the extension period is to allow patients who wish to do so to follow the telemonitoring program until its marketing, regardless of the randomization group on initial inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Men or women patient with heart failure having been hospitalized for cardiac decompensation during the last 12 months.
* Patient with access to a wireline telephone service or GPRS network.
* The patient is willing and able to sign an informed written consent
* Patient is insured under the social security system

Exclusion Criteria:

* No available echocardiographic evaluation.
* BNP lower than 100pg/ml or NT-proBNP lower than 300pg/ml
* A prognosis of a life span of less than 12 months (apart from heart failure)
* Dialysis patients
* Heart transplant or cardiac assist devices
* Patients involved in inotropic treatment
* Patient doesn't have the necessary autonomy to use the equipment
* Patient enrolled in another clinical trial
* A pregnant or nursing woman, or patient of reproductive age who doesn't use contraceptives
* Patients under tutorship, curatorship or judicial protection

Inclusion Criteria in the extension period:

Participation in the open extension period is only offered to patients who participated in the comparative period of the study, did not withdraw prematurely from the latter and gave their free informed written consent to participate to the extension period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 990 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel GALINIER, MD-PhD, Principal Investigator — Rangueil University Hospital - Toulouse; Atul PATHAK, MD-PhD, Principal Investigator — Clinique Pasteur
Locations (38):
- France (37):
  - Cabinet de Cardiologie - Pôle médical spécialisé, Béziers, Languedoc-Rousillon
  - Centre Hospitalier de Béziers, Béziers, Languedoc-Roussillon
  - Cabinet libéral, Saint-Yrieix-la-Perche, Limousin
  - Cabinet libéral de Cardiologie du Muret, Muret, Midi-pyrenées
  - Centre Hospitalier Général d'Auch, Auch, Midi-Pyrénées
  - Centre de réadaptation cardiovasculaire Midi-Gascogne, Beaumont-de-Lomagne, Midi-Pyrénées
  - Centre Hospitalier de Cahors, Cahors, Midi-Pyrénées
  - Centre Hospitalier Intercommunal Castres-Mazamet, Castres, Midi-Pyrénées
  - Clinique des Cèdres, Cornebarrieu, Midi-Pyrénées
  - Clinique de l'Union et du Vaurais, L'Union, Midi-Pyrénées
  - Clinique du Pont de Chaume, Montauban, Midi-Pyrénées
  - Centre Hospitalier de Rodez, Rodez, Midi-Pyrénées
  - Centre Hospitalier Intercommunal du Val d'Ariège, Saint-Jean-de-Verges, Midi-Pyrénées
  - Polyclinique de l'Ormeau, Tarbes, Midi-Pyrénées
  - Centre Hospitalier Universitaire de Toulouse - Hôpital de Rangueil, Toulouse, Midi-Pyrénées
  - Clinique Pasteur, Toulouse, Midi-Pyrénées
  - Hôpital Joseph Ducuing, Toulouse, Midi-Pyrénées
  - Centre Hospitalier Universitaire d'Amiens de Picardie, Amiens
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Centre Hospitalier d'Avignon - Hospital Henri Duffaut, Avignon
  - Centre Hospitalier de Bastia, Bastia
  - Centre Hospitalier Universitaire Bordeaux - Hôpital Saint André, Bordeaux
  - Centre Hospitalier Universitaire de Brest, Brest
  - Centre Hospitalier Universitaire de Lyon - Hôpital Louis Pradel, Bron
  - Centre Hospitalier Universitaire François Mitterrand - Cardiologie 2 : Rythmologie et Insuffisance Cardiaque, Dijon
  - Centre Hospitalier Universitaire François Mitterrand - Cardiologie Générale, Dijon
  - Hôpital Léon Bérard, Hyères
  - Centre Hospitalier Universitaire de Grenoble - Hôpital Antoine Michallon, La Tronche
  - Centre Hospitalier Universitaire de Limoges - Hôpital Dupuytren, Limoges
  - Centre Hospitalier Universitaire de Marseille - Hôpital Nord, Marseille
  - Centre Hospitalier Régional Universitaire de Montpellier, Montpellier
  - Centre Hospitalier Universitaire de Nice - Hôpital Pasteur, Nice
  - Centre Hospitalier Universitaire Caremeau, Nîmes
  - Centre Hospitalier de Pau, Pau
  - Centre Hospitalier Universitaire Bordeaux - Hôpital Haut Lévêque, Pessac
  - Centre Hospitalier de Périgueux, Périgueux
  - Centre Hospitalier Intercommunal de Toulon - La Seyne-sur-Mer, Toulon
- Centre Hospitalier Universitaire de Martinique, Fort-de-France, Martinique

REFERENCES:
- [Result] Galinier M, Roubille F, Berdague P, Brierre G, Cantie P, Dary P, Ferradou JM, Fondard O, Labarre JP, Mansourati J, Picard F, Ricci JE, Salvat M, Tartiere L, Ruidavets JB, Bongard V, Delval C, Lancman G, Pasche H, Ramirez-Gil JF, Pathak A; OSICAT Investigators. Telemonitoring versus standard care in heart failure: a randomised multicentre trial. Eur J Heart Fail. 2020 Jun;22(6):985-994. doi: 10.1002/ejhf.1906. Epub 2020 Jun 15. PMID 32438483

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 13, 2013 and June 22, 2016, 990 patients were enrolled at 38 French centers. Last patient completed 18-month comparative period on December 20, 2017. After this 18-month period, 20 patients entered the non-comparative extension period between June 1, 2017 and March 27, 2018. Last patient completed extension period on September 28, 2018.
Groups:
- Standard Care: * Period 1: Standard follow-up, with conventional monitoring involving consultations and monitoring by their general practitioners or referring cardiologists.
  * Period 2: Patients on standard follow-up during Period 1 were equipped with the Telecardiology Program if they wished and consented to enter the extension period.
- Tele-cardiology Group: Device: Telecardiology Program
  - Period 1: The telecardiology program is a combination of a scale, a device asking the patients questions about the symptoms associated with their heart failure, and regular phone calls made by nurses.
  Automatic algorithms have been built-up in order to detect early the need for a hospitalization due to heart failure.
  - Period 2: Patients on Telecardiology Program during Period 1 were allowed to continue it until its marketing if they wished and consented to enter the extension period.
Period: 18-month Comparative Study Period
Arm/Group | Standard Care | Tele-cardiology Group
Started (990 patients signed an informed consent, 937 returned home and started their ambulatory monitoring. These 937 patients constituted the "Intent to Treat" (ITT) population: 455 patients were in the Standard Care group and 482 patients in the Tele-cardiology Group.) | 455 | 482
Completed | 327 | 305
Not Completed | 128 | 177
Not completed — Death | 90 | 97
Not completed — Withdrawal by Subject | 23 | 52
Not completed — Lost to Follow-up | 6 | 7
Not completed — Heart transplant | 9 | 15
Not completed — Inclusion in another protocol | 0 | 2
Not completed — Hemiplegia | 0 | 1
Not completed — Alzheimer's disease | 0 | 1
Not completed — Move | 0 | 1
Not completed — Hearing loss | 0 | 1
Period: Extension Period
Arm/Group | Standard Care | Tele-cardiology Group
Started | 7 (Standard Care/Tele-cardiology : Patients entered Period 2 if they wished and consented) | 13 (Tele-cardiology/Tele-cardiology : Patients entered Period 2 if they wished and consented)
Completed | 5 | 10
Not Completed | 2 | 3
Not completed — Death | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Heart transplant | 1 | 0
Not completed — Wrong device use | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT population included all study patients randomized once, who left the hospital alive and continued their study participation after their home return and who were not included in the 2 study centers where investigators withdrew their participation.
Groups:
- Tele-cardiology Group: The telecardiology program is a combination of a scale, a device asking the patients questions about the symptoms associated with their heart failure, and regular phone calls made by nurses.
  Automatic algorithms have been built-up in order to detect early the need for a hospitalization due to heart failure.
- Total: Total of all reporting groups
Arm/Group | Standard Care | Tele-cardiology Group | Total
Number analyzed (Participants) | 455 | 482 | 937
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (12.5) | 70.0 (12.4) | 69.9 (12.4)
Age, Customized [Count of Participants; unit: Participants]
  < 60 years | 105 | 93 | 198
  ≥ 60 and < 80 years | 237 | 268 | 505
  ≥ 80 years | 113 | 121 | 234
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 128 | 260
  Male | 323 | 354 | 677
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  France | 455 | 482 | 937
NYHA classification [Count of Participants; unit: Participants] — NYHA: New York Heart Association functional classification categories chronic heart failure patients in 4 stages based on how much they are limited during physical activity. Stage I corresponds to 'No limitation of physical activity', Stage II to 'Slight limitation of physical activity', Stage III to 'Marked limitation of physical activity' and Stage IV to 'Unable to carry on any physical activity without discomfort, symptoms of heart failure at rest Population: Difference from the overall number of baseline participants due to missing data.
  Participants
    number analyzed (Participants) | 452 | 475 | 927
    I | 32 | 29 | 61
    II | 196 | 210 | 406
    III | 185 | 182 | 367
    IV | 39 | 54 | 93
Cardiopathy [Count of Participants; unit: Participants] — Population: Difference from the overall number of baseline participants due to missing data.
  Participants
    number analyzed (Participants) | 454 | 481 | 935
    Ischemic | 211 | 232 | 443
    Non Ischemic | 243 | 249 | 492
Heart failure [Count of Participants; unit: Participants] — Population: Difference from the overall number of baseline participants due to missing data.
  Participants
    number analyzed (Participants) | 453 | 480 | 933
    Left | 184 | 185 | 369
    Right | 34 | 24 | 58
    Global | 235 | 271 | 506
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: Percentage] — Left ventricular ejection fraction refers to the percentage of blood that is pumped out of the filled left ventricle with each contraction of this ventricle. It is calculated on echocardiography mainly. It is the percentage corresponding to the ratio of heart stroke volume (which is the difference between end-diastolic volume and end-systolic volume) divided by end-diastolic volume. Population: Difference from the overall number of baseline participants due to missing data.
  Percentage
    number analyzed (Participants) | 455 | 479 | 934
    (all) | 38.1 (15.2) | 39.3 (14.5) | 38.7 (14.9)
Left Ventricular Ejection Fraction (LVEF), categorical [Count of Participants; unit: Participants] — Population: Difference from the overall number of baseline participants due to missing data.
  Participants
    number analyzed (Participants) | 455 | 479 | 934
    ≤ 40% | 280 | 280 | 560
    > 40% and ≤ 50% | 89 | 95 | 184
    > 50% | 86 | 104 | 190
BNP [Median (Inter-Quartile Range); unit: pg/mL] — BNP: B-type Natriuretic Peptide Population: Difference from the overall number of baseline participants due to missing data and assay of either BNP or NT pro BNP for each participant.
  pg/mL
    number analyzed (Participants) | 191 | 211 | 402
    (all) | 484 [301 to 929] | 510 [303 to 900] | 501 [303 to 911]
NT-pro-BNP [Median (Inter-Quartile Range); unit: pg/mL] — N-Terminal-pro-B-type Natriuretic Peptide Population: Difference from the overall number of baseline participants due to missing data and assay of either NT pro BNP or BNP for each participant.
  pg/mL
    number analyzed (Participants) | 265 | 269 | 534
    (all) | 3277 [1666 to 6914] | 3519 [1778 to 6553] | 3379 [1732 to 6694]
Previous participation in an ETP [Count of Participants; unit: Participants] — ETP= Educational Therapeutic Program
  Participants
    Yes | 114 | 109 | 223
    No | 341 | 373 | 714
Arterial hypertension [Count of Participants; unit: Participants]
  Yes | 246 | 296 | 542
  No | 209 | 186 | 395
Dyslipidemia [Count of Participants; unit: Participants]
  Yes | 248 | 269 | 517
  No | 207 | 213 | 420
Family History of Cardiovascular Disease [Count of Participants; unit: Participants]
  Yes | 73 | 109 | 182
  No | 382 | 373 | 755
Obesity [Count of Participants; unit: Participants] — Obesity defined as Body Mass Index (BMI) ≥ 30.0 kg/m²
  Participants
    Yes | 122 | 140 | 262
    No | 333 | 342 | 675
Smoking [Count of Participants; unit: Participants]
  Yes | 116 | 111 | 227
  No | 339 | 371 | 710
Coronary heart disease [Count of Participants; unit: Participants]
  Yes | 228 | 236 | 464
  No | 227 | 246 | 473
Diabetes mellitus [Count of Participants; unit: Participants]
  Yes | 161 | 146 | 307
  No | 294 | 336 | 630
Chronic renal disease [Count of Participants; unit: Participants] — Population: Difference from the overall number of baseline participants due to missing data.
  Participants
    number analyzed (Participants) | 455 | 481 | 936
    Yes | 128 | 129 | 257
    No | 327 | 352 | 679
Chronic Obstructive Pulmonary Disease [Count of Participants; unit: Participants]
  Yes | 89 | 89 | 178
  No | 366 | 393 | 759
Implantable cardioverter-defibrillator [Count of Participants; unit: Participants]
  Yes | 60 | 60 | 120
  No | 395 | 422 | 817
Cardiac resynchronization therapy [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 1
  No | 454 | 482 | 936
Loop diuretics [Count of Participants; unit: Participants]
  Yes | 417 | 447 | 864
  No | 38 | 35 | 73
Beta-blockers [Count of Participants; unit: Participants]
  Yes | 367 | 379 | 746
  No | 88 | 103 | 191
ACE inhibitors or ARBs [Count of Participants; unit: Participants] — ACE: Angiotensin-Converting Enzyme; ARB: Angiotensin II Receptor Blocker
  Participants
    Yes | 345 | 354 | 699
    No | 110 | 128 | 238
Aldosterone antagonists [Count of Participants; unit: Participants]
  Yes | 211 | 220 | 431
  No | 244 | 262 | 506
Ivabradine [Count of Participants; unit: Participants] — Population: Difference from the overall number of baseline participants due to missing data.
  Participants
    number analyzed (Participants) | 453 | 479 | 932
    Yes | 37 | 23 | 60
    No | 416 | 456 | 872
Digoxin [Count of Participants; unit: Participants] — Population: Difference from the overall number of baseline participants due to missing data.
  Participants
    number analyzed (Participants) | 454 | 481 | 935
    Yes | 15 | 28 | 43
    No | 439 | 453 | 892
Glomerular Filtration Rate (GFR) [Mean (Standard Deviation); unit: mL/min] — Glomerular Filtration Rate estimated using Modification of Diet in Renal Disease (MDRD) formula Population: Difference from the overall number of baseline participants due to missing data.
  mL/min
    number analyzed (Participants) | 455 | 478 | 933
    (all) | 60.6 (25.1) | 60.5 (25.5) | 60.5 (25.3)
Weight [Mean (Standard Deviation); unit: kg] | 77.2 (17.8) | 79.3 (18.2) | 78.3 (18.0)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 27.1 (5.5) | 27.6 (6.0) | 27.4 (5.8)
Supine systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 118.9 (19.3) | 119.6 (19.9) | 119.3 (19.6)
Supine diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 69.5 (12.2) | 69.9 (11.2) | 69.7 (11.7)
Supine pulse rate [Mean (Standard Deviation); unit: beats/min] — Population: Difference from the overall number of baseline participants due to missing data.
  beats/min
    number analyzed (Participants) | 455 | 481 | 936
    (all) | 72.7 (13.9) | 73.7 (15.4) | 73.2 (14.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of All Causes Deaths and (Unplanned) Hospitalizations
Description: Composite morbidity-mortality criterion combining the number of unplanned hospitalizations for any cause and deaths from any cause (adjudicated events)
Time Frame: 18 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Standard Care | Tele-cardiology Group
Number analyzed (Participants) | 455 | 482
Events | 1.46 (1.98) | 1.30 (1.85)
Statistical Analysis 1: Comparison: Standard Care vs Tele-cardiology Group; Number of events compared using a negative binomial regression model with log link for the expected rate of events (i.e., number of events divided by the effective duration of follow-up). Deaths that occurred during hospitalization with an overnight stay were counted as two events; Test type: Superiority; p = 0.80, negative binomial regression; rate ratio = 0.97, 95% CI 2-sided [0.77 to 1.23]

2. Primary Outcome: Number of All Causes Deaths and (Unplanned) Hospitalizations in NYHA Class III or IV Patients
Description: as for outcome 1
Time Frame: 18 months
Population: ITT population with New York Heart Association (NYHA) class III or IV at inclusion (N=460 patients)
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Standard Care | Tele-cardiology Group
Number analyzed (Participants) | 224 | 236
Events | 1.99 (2.26) | 1.53 (1.98)
Statistical Analysis 1: Comparison: Standard Care vs Tele-cardiology Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.18, negative binomial regression; rate ratio = 0.82, 95% CI 2-sided [0.62 to 1.10]

3. Primary Outcome: Number of All Causes Deaths and (Unplanned) Hospitalizations in Socially Isolated Patients
Description: as for outcome 1
Time Frame: 18 months
Population: ITT population with socially isolated status at inclusion (N=216 patients) defined as: either i) SF-36 Mental Health score <45; or ii) Mental Component Summary score <35; or iii) combination of Mental Health score <50 plus Mental Component Summary score <40; or iv) medical history of depression or mood disorders/alterations; or v) use of concomitant antidepressant medications
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Standard Care | Tele-cardiology Group
Number analyzed (Participants) | 104 | 112
Events | 1.89 (2.14) | 1.30 (1.66)
Statistical Analysis 1: Comparison: Standard Care vs Tele-cardiology Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.02, negative binomial regression; rate ratio = 0.60, 95% CI 2-sided [0.39 to 0.92]

4. Secondary Outcome: Time to First Unplanned Hospital Readmission or Death From Any Cause
Description: Time to first unplanned hospital readmission (adjudicated events) or death from any cause, whichever occurred first in the subgroup of patients concerned
Time Frame: 18 months
Population: ITT population
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard Care | Tele-cardiology Group
Number analyzed (Participants) | 254 | 255
days | 84 [29 to 238] | 105 [30 to 232]
Statistical Analysis 1: Comparison: Standard Care vs Tele-cardiology Group; Time to first event compared using the log-rank test; Test type: Superiority; p = 0.68, Log Rank

5. Secondary Outcome: All Causes Deaths - Number of Patients Who Died From Any Cause
Description: Number of patients who died from any cause
Time Frame: 18 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Tele-cardiology Group
Number analyzed (Participants) | 455 | 482
Participants | 89 | 91

6. Secondary Outcome: Time to Death From Any Cause
Description: Time to death from any cause in the subgroup of patients who died
Time Frame: 18 months
Population: ITT population
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard Care | Tele-cardiology Group
Number analyzed (Participants) | 89 | 91
days | 233 [100 to 390] | 252 [148 to 369]
Statistical Analysis 1: Comparison: Standard Care vs Tele-cardiology Group; Time to death from any cause compared using the log-rank test; Test type: Superiority; p = 0.85, Log Rank

7. Secondary Outcome: Number of Unplanned Hospitalizations for Any Cause
Description: Number of unplanned hospitalizations for any cause (adjudicated events)
Time Frame: 18 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Standard Care | Tele-cardiology Group
Number analyzed (Participants) | 455 | 482
Events | 1.27 (1.82) | 1.11 (1.67)
Statistical Analysis 1: Comparison: Standard Care vs Tele-cardiology Group; Number of events compared using a negative binomial regression model with log link for the expected rate of events (i.e., number of events divided by the effective duration of follow-up); Test type: Superiority; p = 0.77, negative binomial regression; rate ratio = 0.97, 95% CI 2-sided [0.78 to 1.21]

8. Secondary Outcome: Number of Deaths and Unplanned Hospitalizations From Cardiovascular Cause
Description: Composite morbidity-mortality criterion combining the number of cardiovascular unplanned hospitalizations and deaths from cardiovascular cause (adjudicated events)
Time Frame: 18 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Standard Care | Tele-cardiology Group
Number analyzed (Participants) | 455 | 482
Events | 1.07 (1.75) | 0.96 (1.56)
Statistical Analysis 1: Comparison: Standard Care vs Tele-cardiology Group; Number of events compared using a negative binomial regression model with log link for the expected rate of events (i.e., number of events divided by the effective duration of follow-up). Deaths from cardiovascular cause that occurred during a hospitalization for cardiovascular cause with an overnight stay were counted as two events; Test type: Superiority; p = 0.83, negative binomial regression; rate ratio = 0.97, 95% CI 2-sided [0.74 to 1.27]

9. Secondary Outcome: Number of Unplanned Hospitalizations for Heart Failure
Description: Number of unplanned hospitalizations for heart failure (adjudicated events)
Time Frame: 18 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Standard Care | Tele-cardiology Group
Number analyzed (Participants) | 455 | 482
Events | 0.75 (1.42) | 0.59 (1.26)
Statistical Analysis 1: Comparison: Standard Care vs Tele-cardiology Group; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.28, negative binomial regression; rate ratio = 0.84, 95% CI 2-sided [0.62 to 1.15]

10. Secondary Outcome: Number of Unplanned Hospitalizations for Heart Failure in NYHA Class III or IV Patients
Description: Number of unplanned hospitalizations for heart failure (adjudicated events)
Time Frame: 18 months
Population: ITT population with New York Heart Association (NYHA) class III or IV at inclusion (N=460 patients)
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Standard Care | Tele-cardiology Group
Number analyzed (Participants) | 224 | 236
Events | 1.02 (1.68) | 0.70 (1.36)
Statistical Analysis 1: Comparison: Standard Care vs Tele-cardiology Group; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.078, negative binomial regression; rate ratio = 0.71, 95% CI 2-sided [0.48 to 1.04]

11. Secondary Outcome: Number of Unplanned Hospitalizations for Heart Failure in Socially Isolated Patients
Description: Number of unplanned hospitalizations for heart failure (adjudicated events)
Time Frame: 18 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Standard Care | Tele-cardiology Group
Number analyzed (Participants) | 104 | 112
Events | 1.00 (1.61) | 0.58 (1.15)
Statistical Analysis 1: Comparison: Standard Care vs Tele-cardiology Group; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.023, negative binomial regression; rate ratio = 0.50, 95% CI 2-sided [0.28 to 0.91]

12. Secondary Outcome: Time to First Unplanned Hospital Readmission for Heart Failure
Description: Time to first unplanned hospital readmission for heart failure (adjudicated events) in the subgroup of patients concerned
Time Frame: 18 months
Population: ITT population
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard Care | Tele-cardiology Group
Number analyzed (Participants) | 160 | 141
days | 79 [28 to 236] | 97 [32 to 252]
Statistical Analysis 1: Comparison: Standard Care vs Tele-cardiology Group; Time to first unplanned hospital readmission for heart failure compared using multivariable Cox regression model; Test type: Superiority; p = 0.044, Regression, Cox; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.62 to 0.99]

13. Secondary Outcome: Evolution of Quality of Life Assessed by Short Form-36 (SF-36) Questionnaire Scores
Description: Evolution of Quality of Life assessed using absolute changes from baseline of each dimension and both component summary scores of SF-36 questionnaire. Indeed, SF-36 questionnaire include 8 general dimensions and 2 composite scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). They are standardized to range between 0 and 100. Higher scores on all SF-36 scales indicate more favorable levels of functioning and less disability. Thus, higher Physical Functioning scores reflect higher physical functioning. Higher Role Physical scores reflect lower limitations due to physical problems. Higher Bodily Pain scores reflect less bodily pain. Higher General Health scores reflect higher general health perception. Higher Vitality scores reflect higher vitality. Higher Social Functioning scores reflect higher social functioning. Higher Role Emotional scores reflect lower limitations due to emotional problems. Higher Mental Health scores reflect better mental health.
Time Frame: Between baseline and 12 months and between baseline and 18 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | Tele-cardiology Group
Number analyzed (Participants) | 323 | 307
score on a scale
  Physical Functioning - 12 months | -1.3 (27.3) | 0.0 (28.0)
  Physical Functioning - 18 months: number analyzed (Participants) | 303 | 284
  Physical Functioning - 18 months | 2.4 (26.3) | 1.3 (28.3)
  Role Physical - 12 Months: number analyzed (Participants) | 322 | 307
  Role Physical - 12 Months | 12.5 (48.0) | 12.5 (48.0)
  Role Physical - 18 Months: number analyzed (Participants) | 303 | 284
  Role Physical - 18 Months | 20.5 (40.2) | 20.7 (41.1)
  Bodily Pain - 12 Months: number analyzed (Participants) | 322 | 307
  Bodily Pain - 12 Months | 1.9 (38.8) | 4.1 (36.9)
  Bodily Pain - 18 Months: number analyzed (Participants) | 303 | 284
  Bodily Pain - 18 Months | 0.6 (35.8) | 4.6 (33.6)
  General Health - 12 Months: number analyzed (Participants) | 321 | 307
  General Health - 12 Months | 0.4 (21.7) | 3.4 (22.3)
  General Health - 18 Months: number analyzed (Participants) | 303 | 284
  General Health - 18 Months | 5.2 (20.4) | 6.8 (22.5)
  Vitality - 12 Months: number analyzed (Participants) | 322 | 307
  Vitality - 12 Months | 5.7 (22.1) | 9.0 (23.7)
  Vitality - 18 Months: number analyzed (Participants) | 303 | 284
  Vitality - 18 Months | 7.3 (21.7) | 11.1 (21.8)
  Social Functioning - 12 Months: number analyzed (Participants) | 321 | 307
  Social Functioning - 12 Months | -0.3 (35.5) | 4.4 (33.8)
  Social Functioning - 18 Months: number analyzed (Participants) | 303 | 284
  Social Functioning - 18 Months | 3.2 (33.3) | 3.8 (33.9)
  Role Emotional - 12 Months: number analyzed (Participants) | 322 | 307
  Role Emotional - 12 Months | -4.3 (45.7) | -2.7 (46.9)
  Role Emotional - 18 Months: number analyzed (Participants) | 302 | 284
  Role Emotional - 18 Months | 6.0 (35.8) | 8.3 (35.9)
  Mental Health - 12 Months: number analyzed (Participants) | 321 | 307
  Mental Health - 12 Months | 1.6 (19.4) | 3.9 (18.8)
  Mental Health - 18 Months: number analyzed (Participants) | 303 | 284
  Mental Health - 18 Months | 3.3 (18.9) | 4.3 (18.5)
  Physical Component Summary - 12 Months: number analyzed (Participants) | 321 | 307
  Physical Component Summary - 12 Months | 1.5 (11.2) | 2.2 (11.1)
  Physical Component Summary - 18 Months: number analyzed (Participants) | 302 | 284
  Physical Component Summary - 18 Months | 2.9 (10.6) | 3.2 (10.7)
  Mental Component Summary - 12 Months: number analyzed (Participants) | 321 | 307
  Mental Component Summary - 12 Months | 0.1 (10.8) | 1.8 (11.3)
  Mental Component Summary - 18 Months: number analyzed (Participants) | 302 | 284
  Mental Component Summary - 18 Months | 2.0 (10.4) | 3.1 (10.4)
Statistical Analysis 1: Comparison: Standard Care vs Tele-cardiology Group; ANCOVA Physical Functioning score: Parametric analysis of covariance mixed model on repeated measurements (Baseline, 12 and 18 months) with physical functioning score assessed at baseline as covariate, study group and visit as fixed factors, interaction between study group and visit, interaction between study group and score assessed at baseline and patient as random factor; Test type: Superiority; p = 0.17, Mixed Models Analysis — Study group effect over time; Adjusted Means Difference = 1.06, 95% CI 2-sided [-2.48 to 4.61]
Statistical Analysis 2: Comparison: Standard Care vs Tele-cardiology Group; ANCOVA Role Physical score: Parametric analysis of covariance mixed model on repeated measurements (Baseline, 12 and 18 months) with role physical score assessed at baseline as covariate, study group and visit as fixed factors, interaction between study group and visit, interaction between study group and score assessed at baseline and patient as random factor; Test type: Superiority; p = 0.23, Mixed Models Analysis — Study group effect over time; Adjusted Means Difference = 1.80, 95% CI 2-sided [-2.61 to 6.21]
Statistical Analysis 3: Comparison: Standard Care vs Tele-cardiology Group; ANCOVA Bodily Pain score: Parametric analysis of covariance mixed model on repeated measurements (Baseline, 12 and 18 months) with bodily pain score assessed at baseline as covariate, study group and visit as fixed factors, interaction between study group and visit, interaction between study group and score assessed at baseline and patient as random factor; Test type: Superiority; p = 0.50, Mixed Models Analysis — Study group effect over time; Adjusted Means Difference = 4.46, 95% CI 2-sided [0.59 to 8.33]
Statistical Analysis 4: Comparison: Standard Care vs Tele-cardiology Group; ANCOVA General Health score: Parametric analysis of covariance mixed model on repeated measurements (Baseline, 12 and 18 months) with general health score assessed at baseline as covariate, study group and visit as fixed factors, interaction between study group and visit, interaction between study group and score assessed at baseline and patient as random factor; Test type: Superiority; p = 0.19, Mixed Models Analysis — Study group effect over time; Adjusted Means Difference = 2.52, 95% CI 2-sided [-0.07 to 5.12]
Statistical Analysis 5: Comparison: Standard Care vs Tele-cardiology Group; ANCOVA Vitality score: Parametric analysis of covariance mixed model on repeated measurements (Baseline, 12 and 18 months) with vitality score assessed at baseline as covariate, study group and visit as fixed factors, interaction between study group and visit, interaction between study group and score assessed at baseline and patient as random factor; Test type: Superiority; p = 0.034, Mixed Models Analysis — Study group effect over time; Adjusted Means Difference = 2.38, 95% CI 2-sided [-0.09 to 4.85]
Statistical Analysis 6: Comparison: Standard Care vs Tele-cardiology Group; ANCOVA Social Functioning score: Parametric analysis of covariance mixed model on repeated measurements (Baseline, 12 and 18 months) with social functioning score assessed at baseline as covariate, study group and visit as fixed factors, interaction between study group and visit, interaction between study group and score assessed at baseline and patient as random factor; Test type: Superiority; p = 0.025, Mixed Models Analysis — Study group effect over time; Adjusted Means Difference = 4.03, 95% CI 2-sided [0.60 to 7.47]
Statistical Analysis 7: Comparison: Standard Care vs Tele-cardiology Group; ANCOVA Role Emotional score: Parametric analysis of covariance mixed model on repeated measurements (Baseline, 12 and 18 months) with role emotional score assessed at baseline as covariate, study group and visit as fixed factors, interaction between study group and visit, interaction between study group and score assessed at baseline and patient as random factor; Test type: Superiority; p = 0.90, Mixed Models Analysis — Study group effect over time; Adjusted Means Difference = 1.01, 95% CI 2-sided [-2.79 to 4.81]
Statistical Analysis 8: Comparison: Standard Care vs Tele-cardiology Group; ANCOVA Mental Health score: Parametric analysis of covariance mixed model on repeated measurements (Baseline, 12 and 18 months) with mental health score assessed at baseline as covariate, study group and visit as fixed factors, interaction between study group and visit, interaction between study group and score assessed at baseline and patient as random factor; Test type: Superiority; p = 0.19, Mixed Models Analysis — Study group effect over time; Adjusted Means Difference = 2.26, 95% CI 2-sided [0.16 to 4.37]
Statistical Analysis 9: Comparison: Standard Care vs Tele-cardiology Group; ANCOVA Physical Component Summary (PCS) score: Parametric analysis of covariance mixed model on repeated measurements (Baseline, 12 and 18 months) with PCS score assessed at baseline as covariate, study group and visit as fixed factors, interaction between study group and visit, interaction between study group and score assessed at baseline and patient as random factor; Test type: Superiority; p = 0.26, Mixed Models Analysis — Study group effect over time; Adjusted Means Difference = 0.90, 95% CI 2-sided [-0.48 to 2.28]
Statistical Analysis 10: Comparison: Standard Care vs Tele-cardiology Group; ANCOVA Mental Component Summary (MCS) score: Parametric analysis of covariance mixed model on repeated measurements (Baseline, 12 and 18 months) with MCS score assessed at baseline as covariate, study group and visit as fixed factors, interaction between study group and visit, interaction between study group and score assessed at baseline and patient as random factor; Test type: Superiority; p = 0.17, Mixed Models Analysis — Study group effect over time; Adjusted Means Difference = 1.20, 95% CI 2-sided [0.08 to 2.31]

14. Secondary Outcome: Annualized Number of Unplanned Hospitalizations for Any Cause During the Extension Period
Description: Annualized number of unplanned hospitalizations for any cause according to investigators in patients hospitalized at least once during the extension period
Time Frame: Extension period until the marketing of the telemonitoring program (from 2 to 16 months, with an average of 9.5 months)
Population: Extension Period Set
Measure: Mean (Standard Deviation); unit: Events
Groups:
- Standard Care/Tele-cardiology: * Period 1: Standard follow-up, with conventional monitoring involving consultations and monitoring by their general practitioners or referring cardiologists.
  * Period 2: Patients on standard follow-up during Period 1 were equipped with the Telecardiology Program if they wished and consented to enter the extension period.
- Tele-cardiology/Tele-cardiology: - Period 1: The telecardiology program is a combination of a scale, a device asking the patients questions about the symptoms associated with their heart failure, and regular phone calls made by nurses.
  Automatic algorithms have been built-up in order to detect early the need for a hospitalization due to heart failure.
  - Period 2: Patients on Telecardiology Program during Period 1 were allowed to continue it until its marketing if they wished and consented to enter the extension period.
Arm/Group | Standard Care/Tele-cardiology | Tele-cardiology/Tele-cardiology
Number analyzed (Participants) | 2 | 5
Events | 1.30 (0.57) | 3.30 (2.09)

15. Secondary Outcome: Number of Patients Who Died From Any Cause During the Extension Period
Description: Number of patients who died from any cause during the extension period
Time Frame: Extension period until the marketing of the telemonitoring program (from 2 to 16 months, with an average of 9.5 months)
Population: Extension Period Set
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care/Tele-cardiology | Tele-cardiology/Tele-cardiology
Number analyzed (Participants) | 7 | 13
Participants | 0 | 2

16. Secondary Outcome: Annualized Number of Unplanned Hospitalizations From Cardiovascular Cause During the Extension Period
Description: Annualized number of unplanned hospitalizations from cardiovascular cause according to investigators in patients hospitalized at least once for cardiovascular cause during the extension period
Time Frame: Extension period until the marketing of the telemonitoring program (from 2 to 16 months, with an average of 9.5 months)
Population: Extension Period Set
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Standard Care/Tele-cardiology | Tele-cardiology/Tele-cardiology
Number analyzed (Participants) | 2 | 5
Events | 1.30 (0.57) | 2.84 (1.18)

17. Secondary Outcome: Number of Patients Who Died From Cardiovascular Cause During the Extension Period
Description: Number of patients who died from cardiovascular cause according to investigators during the extension period
Time Frame: Extension period until the marketing of the telemonitoring program (from 2 to 16 months, with an average of 9.5 months)
Population: Extension Period Set
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care/Tele-cardiology | Tele-cardiology/Tele-cardiology
Number analyzed (Participants) | 7 | 13
Participants | 0 | 0

18. Post Hoc Outcome: Time to First Unplanned Hospital Readmission or Death From Any Cause in NYHA Class III or IV Patients
Description: as for outcome 4
Time Frame: 18 months
Population: New York Heart Association (NYHA) class III or IV at inclusion patients with unplanned hospital readmission or death from any cause included in the Overall Number of Participants Analyzed
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard Care | Tele-cardiology Group
Number analyzed (Participants) | 157 | 140
days | 67 [27 to 191] | 82 [29 to 158]
Statistical Analysis 1: Comparison: Standard Care vs Tele-cardiology Group; Time to first event compared using the log-rank test; Test type: Superiority; p = 0.03, Log Rank

19. Post Hoc Outcome: Time to First Unplanned Hospital Readmission or Death From Any Cause in Socially Isolated Patients
Description: as for outcome 4
Time Frame: 18 months
Population: Patients with socially isolated status at inclusion defined as: either i) SF-36 Mental Health score <45; or ii) Mental Component Summary score <35; or iii) combination of Mental Health score <50 plus Mental Component Summary score <40; or iv) medical history of depression or mood disorders/alterations; or v) use of concomitant antidepressant medications and with unplanned hospital readmission or death from any cause included in the Overall Number of Participants Analyzed'
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard Care | Tele-cardiology Group
Number analyzed (Participants) | 70 | 64
days | 81 [28 to 240] | 91 [32 to 277]
Statistical Analysis 1: Comparison: Standard Care vs Tele-cardiology Group; Time to first event compared using the log-rank test; Test type: Superiority; p = 0.15, Log Rank

20. Post Hoc Outcome: Time to First Unplanned Hospital Readmission for Heart Failure in NYHA Class III or IV Patients
Description: as for outcome 12
Time Frame: 18 months
Population: New York Heart Association (NYHA) class III or IV at inclusion patients with unplanned hospital readmission for heart failure included in the Overall Number of Participants Analyzed
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard Care | Tele-cardiology Group
Number analyzed (Participants) | 101 | 78
days | 62 [24 to 182] | 82 [30 to 183]
Statistical Analysis 1: Comparison: Standard Care vs Tele-cardiology Group; Time to first unplanned hospital readmission for heart failure compared using multivariable Cox regression model; Test type: Superiority; p = 0.02, Regression, Cox; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.53 to 0.95]

21. Post Hoc Outcome: Time to First Unplanned Hospital Readmission for Heart Failure in Socially Isolated Patients
Description: as for outcome 12
Time Frame: 18 months
Population: Patients with socially isolated status at inclusion defined as: either i) SF-36 Mental Health score <45; or ii) Mental Component Summary score <35; or iii) combination of Mental Health score <50 plus Mental Component Summary score <40; or iv) medical history of depression or mood disorders/alterations; or v) use of concomitant antidepressant medications and with unplanned hospital readmission for heart failure included in the Overall Number of Participants Analyzed'
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard Care | Tele-cardiology Group
Number analyzed (Participants) | 47 | 31
days | 77 [27 to 231] | 80 [23 to 318]
Statistical Analysis 1: Comparison: Standard Care vs Tele-cardiology Group; Time to first unplanned hospital readmission for heart failure compared using multivariable Cox regression model; Test type: Superiority; p = 0.043, Regression, Cox; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.39 to 0.98]

ADVERSE EVENTS:
Time Frame: During their study participation, patients were only examined once by the investigating cardiologists at the study centers, at the time of their enrolment and randomization. After this Inclusion Visit, patients were followed up via four telephone calls, conducted by clinical study technicians (at 15 days, 6, 12 and 18 months, all ±15 days).
Description: Serious and Other [Not Including Serious] Adverse Events were not monitored/assessed in this study which did not involve any investigational medicinal product.
  Deaths and hospitalizations constituted the study outcome measures and efficacy criteria. Therefore, they were not considered a result from an Adverse Event and were not reported as Serious Adverse Events.
Groups:
- Tele-cardiology Group/Tele-cardiology: - Period 1: The telecardiology program is a combination of a scale, a device asking the patients questions about the symptoms associated with their heart failure, and regular phone calls made by nurses.
  Automatic algorithms have been built-up in order to detect early the need for a hospitalization due to heart failure.
  - Period 2: Patients on Telecardiology Program during Period 1 were allowed to continue it until its marketing if they wished and consented to enter the extension period.
Arm/Group | Standard Care/Tele-cardiology | Tele-cardiology Group/Tele-cardiology
All-Cause Mortality (participants affected / at risk) | 90/455 | 99/482
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
There is no significant methodological limitation in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release, can require changes to the communication and can embargo communications regarding trial results for a period that is less than or equal to 180 days from the time submitted to the sponsor for review. The modifications made by the sponsor cannot in any way affect the scientific value of the publication.

DOCUMENTS (2):
  • Study Protocol (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT02068118/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT02068118/SAP_001.pdf